CLINICAL TRIAL: NCT01899287
Title: A Randomised Clinical Trial on the Effect of Group Education on Skin-protective Behaviour Versus Treatment as Usual Among Individuals With Newly Notified Occupational Hand Eczema
Brief Title: A Randomised Clinical Trial on the Effect of Group Education on Patients With Occupational Hand Eczema
Acronym: PREVEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Tove Agner, professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-1-2012-053
Record Dates: First submitted 2013-07-04; First posted 2013-07-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Eczema; Skin Conditions
Keywords: workers education; occupational
MeSH Terms: conditions — Eczema; Skin Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- education in skin care (Experimental): The experimental intervention consists of:
  A. Group education on general skin-protective behaviour. B. Group education and counselling on work-related skin-protective behaviour, which might extend to a work-place visit.
  C. Social guidance related to OHE. D. Telephone hot-line for work and case-related problems, maintained by nurse.
  Interventions: Behavioral: group education
- no intervention (No Intervention): The control group will not have access to the group education, the profession specific information and the social guidance or the telephone hotline.

INTERVENTIONS:
Behavioral: group education — The experimental intervention consists of:
  A. Group education on general skin-protective behaviour. B. Group education and counselling on work-related skin-protective behaviour, which might extend to a work-place visit.
  C. Social guidance related to OHE. D. Telephone hot-line for work and case-related problems, maintained by nurse.
  Arms: education in skin care

SUMMARY:
Occupational hand eczema (OHE) is a frequent disease which often takes a chronic course. The burden of the disease is high in a personal as well as in a socio-economic context. There is a need for evaluating new strategies to improve the prognosis for OHE patients. The objectives of the study is to evaluate the effect of group education on sick lave, health-related quality of life and disease severity among individuals with newly notified OHE.

The trial population consist of individuals from the Capital Region of Denmark and Region Zealand with a suspected skin-related industrial injury notified to the Danish National Board of Industrial Injuries (DNBII). Recruitment is started Juli 2012, and will continue until the designed number of participants have been included.

All participants will be assessed in a questionnaire at time T=0 with regard to: self evaluated disease severity, health-related quality of life, skin protective behaviour, knowledge of skin protection, self-efficacy, work-role function and if active in workforce. The participants will then be randomised. The intervention group will be invited to participate in the educative course, and work place visits will be offered. In the intervention group a telephone hot line will be available for further questions concerning these topics. The control group will not have access to any of these interventions. Both intervention group and control group will be contacted every eighth week about number of days of sick leave/absence from workforce. Both groups are re-assessed using a questionnaire at T=12 months. There will be a total of 742 included participants.

.

DETAILED DESCRIPTION:
The hypotheses of the PREVEX trial are:

* Early information build on evidence-based skin-protection programmes and work-place visits with counselling in skin care, followed by telephone hotline, will give the participants increased level of knowledge concerning the treatment and prevention of OHE.
* Increased level of knowledge concerning prevention and focus on skin care will have a positive impact on skin-protective behaviour and will lower the severity of HE and prevent the development of chronic eczema.
* The decrease in severity of HE will decrease sick leave and keep the participants in job, or prevent job loss, or facilitate the re-entry into the workforce.
* In total, the intervention will have a positive effect on health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported HE, i.e., individuals answering 'yes' in the questionnaire to the question 'Have you or have you had hand eczema?'
* The questionnaire is sufficiently filled in with respect to 'severity of HE' and 'profession'.
* Written informed consent.

Exclusion Criteria:

* Age below 18 years or above 65 years.
* Permanently excluded from the workforce.
* Inability to understand the Danish language sufficiently to benefit from the course.
* Any serious medical condition which, in the opinion of the investigator, may interfere with the evaluation of the results.
* Lack of written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Sick leave | 1 year
  • Total sick leave; measured as self-reported number of days with sick leave during the trial period.
Health-related quality of life | 1 year
  Health-related quality of life; measured as points scored in the Dermatology Life Quality Index (DLQI) at 12 months after inclusion.
  •
Disease severity | 1 year
  Subjective assessment of hand eczema severity; measured by use of a photographic guide at 12 months after inclusion.

SECONDARY OUTCOMES:
eczema-related sick leave | 1 year
  The following outcomes will be assessed as explorative, as there is insufficient information to conduct power calculations.
  * Eczema-related sick leave; measured as self-reported number of days with eczema-related sick leave during the trial period.
  * Absence registered by the DREAM-register; only absence for more than 28 days from workplace is registered here. This will be done at T=12 months. We will measure absence from work because of sick leave for more than 21 days , yes or no.
  * Behaviour measured as number of points achieved in a questionnaire concerning both occupational and private risk behaviour at time T=12.
  * Knowledge of skin protection measured as numbers of points achieved in a multiple choice questionnaire at time T=12 months.
  * Performance management at time T=12 months of the participant measured by the number of points achieved in:
    * Self-efficacy; and
    * Self-evaluated ability to self-care.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Fisker MH, Agner T, Lindschou J, Bonde JP, Ibler KS, Gluud C, Winkel P, Ebbehoj NE. Protocol for a randomised trial on the effect of group education on skin-protective behaviour versus treatment as usual among individuals with newly notified occupational hand eczema - the Prevention of Hand Eczema (PREVEX) Trial. BMC Dermatol. 2013 Nov 19;13:16. doi: 10.1186/1471-5945-13-16. PMID 24245553